CLINICAL TRIAL: NCT05695105
Title: Novel Treatment for Dental Ankylosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Wei Huang, DMD, PhD, MSD, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro2020003227
Record Dates: First submitted 2022-10-04; First posted 2023-01-23 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Dental Ankylosis
Keywords: Dental ankylosis; Vibration; Electric toothbrush; Mini-implant; Heavy force
MeSH Terms: conditions — Tooth Ankylosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Vibration Group (Experimental): For primary and permanent teeth that will receive only toothbrush vibration treatment.
  Interventions: Device: Electric Toothbrush-Generated Vibration
- Vibration and Mini-implant Group (Experimental): For permanent teeth that will receive mini-implant treatment followed by failed toothbrush vibration treatment.
  Interventions: Device: Electric Toothbrush-Generated Vibration; Device: Mini-Implant-Assisted Orthodontic Treatment

INTERVENTIONS:
Device: Electric Toothbrush-Generated Vibration — Testing electric toothbrush handle-generated vibration to treat ankylosis of teeth
Device: Mini-Implant-Assisted Orthodontic Treatment — Testing mini-implant-assisted heavy force application to treat ankylosis of teeth
  Arms: Vibration and Mini-implant Group

SUMMARY:
The study is to determine whether one (or two) new method(s) will help treat dental ankylosis. This study tackles the challenging tooth-bone fusion disorder of ankylosis. In growing patients, ankylosis causes significant developmental bone defects due to its inhibition of the vertical growth of the affected alveolar bone area.

DETAILED DESCRIPTION:
Currently, there is no treatment available to reverse ankylosis' pathology and therefore it often leads to extraction of the tooth in young patients to prevent more serious pathological complications. In this study, the investigators will use toothbrush-generated vibration and mini-implant-assisted heavy force delivery approaches to treating ankylosis in deciduous and permanent teeth. If successful, the techniques will completely restore the full eruption capacity of an ankylosed tooth by reversing its pathological development. The purpose of the research is to investigate whether a new treatment approach provides an effective noninvasive or minimally invasive treatment for dental ankylosis.

Study participants will be asked to use an electric toothbrush handle to vibrate the ankylosed tooth for 15-60 seconds every day for five days and have a few follow-up visits to the clinic. If the ankylosed tooth is a permanent tooth and the electric toothbrush vibration approach does not work, the participants will be asked to have a six-week period of orthodontic treatment for the tooth with the placement of a mini-implant near the tooth and then have monthly follow-up visits for up to five months.

ELIGIBILITY:
Inclusion Criteria:

* Full informed consent and/or informed assent (minors)
* Be willing and able to comply with all study requirements
* Male or female
* Aged 6-30
* Clinically diagnosed to have either an ankylosed deciduous tooth or a non-third molar mildly- to moderately- ankylosed permanent tooth, and with crown partially visible in the oral cavity. Clinical diagnosis of ankylosis includes the following factors: dental trauma history, infra-eruption with no apparent mechanical obstruction or other cause, contralateral tooth in occlusal contact for over one year, decreased alveolar bone height, no or reduced tooth mobility, and x-ray or cone-beam computer tomography (CBCT) imaging indications of an obliterated PDL space. Ultimately, the diagnosis will be confirmed by lack of tooth movement discovered during orthodontic treatment or when subjected to a heavy force through our study (Phelan M K, et al. 1990).
* English speaking (primary language or fluent)

Exclusion Criteria:

* Severe and extensive ankylosis of permanent teeth as diagnosed through CBCT
* Primary failure of eruption with previous orthodontic treatment
* Any systemic disorders particularly those affecting bleeding or skeletal health
* Any systemic medications
* Any mental or developmental disorders that affect patient understanding or compliance
* Allergic to our local anesthetic drug
* Can pass an infectious disease to someone else right now (e.g., having a flu)
* Is pregnant
* Has a history of smoking
* Have not reached the age of 6 or older than age of 30
* Not cooperative enough during dental examinations
* The dentist finds out that he/she is not able to keep the mini-implant, the brackets and the wires in place around the tooth that is being treated
* Not fluent in English

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
Change from the Baseline Ankylosed Tooth Position During 9 Months Period | For vibration group, it will be on Day 0, 33, 61, 89 if necessary after vibration; for vibration and mini-implant group, it will be on Day 0, 33, 61, 89, 131, 159, 187, 215, 243, 271 if necessary after mini-implant placement.
  The change of ankylosed tooth position will be assessed clinically and radiographically through measuring the distance (mm) of the lowest (maxillary arch) or highest (mandibular arch) cusp tip to the occlusal plane where full occlusal contact would have been established.
Change from the Baseline Alveolar Bone Defect Level of the Ankylosed Tooth During 9 Months Period | For vibration group, it will be on Day 0 and the last day of visit (Day 33, 61 or 89, depending on the outcome); for vibration and mini-implant group, it will be on Day 0 and the last day of visit from the vibration phase and Day 131, 215 if necessary.
  The vertical alveolar bone defect at the ankylosed tooth position will be assessed clinically through measuring the periodontal probing depth (mm) and radiographically through measuring the distance between the alveolar bone attachment position to the neighboring tooth's cementum-enamel junction (CEJ) in the tooth's long axis direction (mm). The change of these measurements will be recorded.

SECONDARY OUTCOMES:
Mobility of Ankylosed Tooth | For vibration group, on Day 0, 6, 33, 61, 89 if necessary; for vibration and mini-implant group on Day 0, 42, 70, 98, 126, 154, 198 if necessary
  The mobility of the ankylosed tooth will be assessed clinically. Mobility will be classified into three Grades:
  Grade 1: < 1 mm (horizontal) Grade 2: > 1 mm (horizontal) Grade 3: > 1 mm (horizontal+vertical mobility)
Ankylosed Tooth Periodontal Ligament (PDL) Obliteration | For vibration and mini-implant group only, on Day 0 and last day of clinical exam (either Day 98, 126, 154, or 198)
  The PDL obliteration will be assessed radiographically using small field of view Cone Bean Computed Tomography (CBCT) images. Examiner will assess the CBCT images and determine the PDL obliteration area and changes (increased, decreased, disappeared).

CONTACTS AND LOCATIONS:
Overall Officials: Wei Huang, DDS, PhD, Principal Investigator — Rutgers School of Dental Medicine
Locations (1):
- Rutgers School of Dental Medicine, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Souza RF, Travess H, Newton T, Marchesan MA. Interventions for treating traumatised ankylosed permanent front teeth. Cochrane Database Syst Rev. 2015 Dec 16;2015(12):CD007820. doi: 10.1002/14651858.CD007820.pub3. PMID 26677103
- [Background] Tieu LD, Walker SL, Major MP, Flores-Mir C. Management of ankylosed primary molars with premolar successors: a systematic review. J Am Dent Assoc. 2013 Jun;144(6):602-11. doi: 10.14219/jada.archive.2013.0171. PMID 23729457
- [Background] Andersson L, Malmgren B. The problem of dentoalveolar ankylosis and subsequent replacement resorption in the growing patient. Aust Endod J. 1999 Aug;25(2):57-61. doi: 10.1111/j.1747-4477.1999.tb00088.x. PMID 11411080
- [Background] Mueller CT, Gellin ME, Kaplan AL, Bohannan HM. Prevalence of ankylosis of primary molars in different regions of the United States. ASDC J Dent Child. 1983 May-Jun;50(3):213-8. No abstract available. PMID 6575989
- [Background] Andersson L, Blomlof L, Lindskog S, Feiglin B, Hammarstrom L. Tooth ankylosis. Clinical, radiographic and histological assessments. Int J Oral Surg. 1984 Oct;13(5):423-31. doi: 10.1016/s0300-9785(84)80069-1. PMID 6438004
- [Background] Oh NY, Nam SH, Lee JS, Kim HJ. Delayed Spontaneous Eruption of Severely Infraoccluded Primary Second Molar: Two Case Reports. J Clin Pediatr Dent. 2020;44(3):185-189. doi: 10.17796/1053-4625-44.3.9. PMID 32644898
- [Background] Djemal S, Karki T, Mack G. Challenges in treating traumatically intruded and ankylosed permanent incisors: a case report with a multidisciplinary approach. Dent Update. 2015 Jan-Feb;42(1):44-6, 49-50. doi: 10.12968/denu.2015.42.1.44. PMID 26062278
- [Background] Mistry VN, Barker CS, James Spencer R. The first permanent molar: spontaneous eruption after a five-year failure. Int J Paediatr Dent. 2017 Sep;27(5):428-433. doi: 10.1111/ipd.12293. Epub 2017 Mar 1. PMID 28247574